CLINICAL TRIAL: NCT04628949
Title: A Single-Use Duodenoscope in a Real-World Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ambu A/S (Industry)
Collaborators: Ambu Inc. (Industry); Infinite Clinical Solutions (Unknown); Prelude Dynamics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIS-018
Record Dates: First submitted 2020-11-05; First posted 2020-11-16 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography (ERCP)
Keywords: Endoscopic Retrograde Cholangiopancreatography; ERCP; Duodenoscope; Endoscope; aScope Duodeno; aBox

STUDY DESIGN:
Intervention Model Description: Prospective, Non-Randomized, Single-Arm, Post-Market Observational Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- aScope™ Duodeno endoscope and aBox™ Duodeno (Experimental): Eligible subjects who are undergoing non-emergent, clinically indicated ERCP using aScope™ Duodeno endoscope and aBox™ Duodeno.
  Interventions: Device: aScope™ Duodeno endoscope and aBox™ Duodeno

INTERVENTIONS:
Device: aScope™ Duodeno endoscope and aBox™ Duodeno — The aScope™ Duodeno endoscope is a sterile single-use disposable duodenoscope indicated for endoscopic retrograde cholangiopancreatography (ERCP) procedures.The aScope™ Duodeno endoscope is designed to be used with aBox Duodeno, endoscopic accessories and other ancillary equipment for ERCP procedures.
  The aBox Duodeno is the console that is necessary for processing the endoscope camera´s video image, regarding the remote switches and output video and recorder data. The aBox Duodeno is designed to be used with the aScope™ Duodeno endoscope.

SUMMARY:
This study will assess how the aScope™ Duodeno endoscope performs in procedures that treat problems of the bile and pancreatic ducts.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single-arm post-market observational clinical study that will assess the single-use Ambu® aScope™ Duodeno for non-emergent, standard of care (SOC) ERCP procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old.
2. Subject is indicated and scheduled for an elective, non-emergent ERCP.
3. Subject is willing and able to give informed consent and HIPAA authorization.

Exclusion Criteria:

1. Subject has altered pancreaticobiliary anatomy including:

   1. Billroth II
   2. Roux-en-Y gastric bypass
   3. Loop gastric bypass
   4. Post-Whipple
   5. Roux-en-Y hepaticojejunostomy
2. Subject requires an emergency ERCP (emergent decompression procedure within 6-12 hours of presentation to prevent life-threatening sequelae).
3. Subject has any of the following severe co-morbid conditions

   1. Morbid obesity (BMI ≥ 40)
   2. Unstable cardiopulmonary conditions
   3. Severe and uncorrectable coagulopathy
   4. Severe and uncorrectable thrombocytopenia
4. Subject has clinically significant esophageal, pyloric or duodenal strictures.
5. Subject has been previously been treated under this investigational plan.
6. Subject is pregnant or female with reproductive capability who is unwilling to have a pre-procedure pregnancy test and use birth control.
7. Subject is actively taking an anticoagulant or antiplatelet agent other than aspirin.
8. Subject, in the opinion of the Investigator, has a severe comorbidity, poor general physical/mental health and/or a condition that will not allow the subject to be a good study candidate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
To evaluate the ERCP procedural success rates with the aScope™ Duodeno endoscope when completing the ERCP procedure for the intended indication(s). | Procedure Completion (Day 0)
  Procedure success will be defined as the successful completion of the ERCP procedure with the aScope™ Duodeno endoscope. The procedural success rate will be the incidence rate of success for the ERCP procedure.

SECONDARY OUTCOMES:
To establish comprehensive performance attributes of aScope™ Duodeno endoscope through its use by multiple endoscopists in conducting various ERCP procedures. | Procedure Completion (Day 0)
  Procedure success for sub categories of ERCP procedures will be defined as the successful completion of the ERCP procedure with the aScope™ Duodeno endoscope. The procedural success rate will be the incidence rate of success for the stratified sub-categories of ERCP procedures with the the aScope™ Duodeno endoscope.
To evaluate rate of conversion to a reusable endoscope, other endoscope or an open procedure from the aScope™ Duodeno endoscope during the ERCP procedure. | Procedure Completion (Day 0)
  Rate of conversion will be measured by the incidence rate of when a conversion to a different endoscope or open procedure is necessitated during the ERCP procedure with the aScope™ Duodeno endoscope.
To evaluate rate of successful completion of a converted ERCP procedure. | Procedure Completion (Day 0)
  Successful completion will be measured by the incidence rate of success for converted ERCP procedure as stratified by the conversion method (reusable scope, other endoscope, other procedure).
To evaluate the device deficiency rate for the aScope™ Duodeno endoscope. | Procedure Completion (Day 0)
  Incidence rate of device deficiencies as defined as either a device failure or device malfunction for the aScope™ Duodeno endoscope during ERCP procedure.
To evaluate physician satisfaction with the aScope™ Duodeno endoscope. | Procedure Completion (Day 0)
  Physician reported outcomes questionnaire on physician satisfaction with the aScope™ Duodeno endoscope for ERCP procedures.

OTHER OUTCOMES:
To evaluate safety of the aScope™ Duodeno endoscope in ERCP. | Day 30 (+3) Post-Procedure
  Safety will be assessed based on the incidence rates of adverse events based on the seriousness and relatedness to the device and/or procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Smith, Study Director — Ambu Inc.
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Colorado Hospital, Aurora, Colorado
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Indiana University, University Hospital, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Mount Sinai South Nassau, Oceanside, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domagk D, Oppong KW, Aabakken L, Czako L, Gyokeres T, Manes G, Meier P, Poley JW, Ponchon T, Tringali A, Bellisario C, Minozzi S, Senore C, Bennett C, Bretthauer M, Hassan C, Kaminski MF, Dinis-Ribeiro M, Rees CJ, Spada C, Valori R, Bisschops R, Rutter MD. Performance measures for endoscopic retrograde cholangiopancreatography and endoscopic ultrasound: A European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. United European Gastroenterol J. 2018 Dec;6(10):1448-1460. doi: 10.1177/2050640618808157. Epub 2018 Oct 19. PMID 30574315
- [Background] Baron, Kozarek, Carr-Locke, et al. ERCP 3rd Edition. Elsevier. 2019.
- [Background] Lee DH, Kim DB, Kim HY, Baek HS, Kwon SY, Lee MH, Park JC. Increasing potential risks of contamination from repetitive use of endoscope. Am J Infect Control. 2015 May 1;43(5):e13-7. doi: 10.1016/j.ajic.2015.01.017. Epub 2015 Feb 25. PMID 25726130
- [Background] Alfa MJ, Olson N, DeGagne P, Jackson M. A survey of reprocessing methods, residual viable bioburden, and soil levels in patient-ready endoscopic retrograde choliangiopancreatography duodenoscopes used in Canadian centers. Infect Control Hosp Epidemiol. 2002 Apr;23(4):198-206. doi: 10.1086/502035. PMID 12002234
- [Background] Petersen BT. Duodenoscope reprocessing: risk and options coming into view. Gastrointest Endosc. 2015 Sep;82(3):484-7. doi: 10.1016/j.gie.2015.07.004. No abstract available. PMID 26279349
- [Background] Ross AS, Baliga C, Verma P, Duchin J, Gluck M. A quarantine process for the resolution of duodenoscope-associated transmission of multidrug-resistant Escherichia coli. Gastrointest Endosc. 2015 Sep;82(3):477-83. doi: 10.1016/j.gie.2015.04.036. Epub 2015 Jun 16. PMID 26092616
- [Background] USA FDA: Medical Device Safety: Safety Communications. The FDA Continues to Remind Facilities of the Importance of Following Duodenoscope Reprocessing Instructions: FDA Safety Communication. 12 April 2019.
- [Background] USA FDA: Medical Device Safety: Safety Communications. The FDA is Recommending Transition to Duodenoscopes with Innovative Designs to Enhance Safety: FDA Safety Communication. 29 August 2019.
- [Background] Balan GG, Rosca I, Ursu EL, Fifere A, Varganici CD, Doroftei F, Turin-Moleavin IA, Sandru V, Constantinescu G, Timofte D, Stefanescu G, Trifan A, Sfarti CV. Duodenoscope-Associated Infections beyond the Elevator Channel: Alternative Causes for Difficult Reprocessing. Molecules. 2019 Jun 25;24(12):2343. doi: 10.3390/molecules24122343. PMID 31242689
- [Background] Cotton PB, Eisen G, Romagnuolo J, Vargo J, Baron T, Tarnasky P, Schutz S, Jacobson B, Bott C, Petersen B. Grading the complexity of endoscopic procedures: results of an ASGE working party. Gastrointest Endosc. 2011 May;73(5):868-74. doi: 10.1016/j.gie.2010.12.036. Epub 2011 Mar 5. PMID 21377673
- [Background] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Background] ASGE Standards of Practice Committee; Chandrasekhara V, Khashab MA, Muthusamy VR, Acosta RD, Agrawal D, Bruining DH, Eloubeidi MA, Fanelli RD, Faulx AL, Gurudu SR, Kothari S, Lightdale JR, Qumseya BJ, Shaukat A, Wang A, Wani SB, Yang J, DeWitt JM. Adverse events associated with ERCP. Gastrointest Endosc. 2017 Jan;85(1):32-47. doi: 10.1016/j.gie.2016.06.051. Epub 2016 Aug 18. No abstract available. PMID 27546389